CLINICAL TRIAL: NCT02269228
Title: Tolerability of a Two Week Treatment With Asasantin Extended Release 200/25 mg Capsules b.i.d., Compared to Reduced Dose During the First Week of Treatment in a Double-blind, Randomised, Placebo Controlled Parallel Group Comparison Trial in Healthy Female and Male Subjects
Brief Title: Tolerability of Asasantin in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9.131
Record Dates: First submitted 2014-10-20; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (3):
- Asasantin ER (Experimental): Administered once daily (days 1 to 7), followed by twice daily administration (days 8 to 14)
  Interventions: Drug: Asasantin ER
- Asasantin ER, administered twice daily from day 1 to day 14 (Experimental)
  Interventions: Drug: Asasantin ER
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asasantin ER
  Arms: Asasantin ER; Asasantin ER, administered twice daily from day 1 to day 14
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate the occurrence of dipyridamole associated headaches in healthy subjects using a titration scheme or not

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy females/males, range from 18 to 55 years of age and be within a Broca Index of ≥ - 20 % and ≤ + 20 %
* Prior to admission to the study all subjects will have given, in accordance with good clinical practice (GCP) and the local legislation, their written informed consent.

Exclusion Criteria:

* Subjects will be excluded from the study if the results of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and are of clinical relevance
* Subjects with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Subjects with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders or neurological disorders
* Subjects with known history of orthostatic hypotension, fainting spells or blackouts
* Subjects with chronic or relevant acute infections
* Subjects with history of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Subjects who have taken a drug with a long half-life (> 24 hours) (≤ 1 month prior to administration or during the trial)
* Subjects who received any other drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Subjects who have participated in another study with an investigational drug (≤ 1 month prior to administration or during the trial)
* Subjects who smoke more than 15 cigarettes or 4 cigars or 4 pipes/day
* Subjects who are not able to refrain from excessive consumption of methylxanthine containing drinks or food
* Subjects who drink more than 60 g of alcohol per day
* Subjects who are dependent on drugs
* Subjects who have donated blood (> 400 ml) (≤ 4 weeks prior to administration or during the trial)
* Subjects who have participated in excessive physical activities (≤ 5 days prior to administration or during the trial)

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (acceptable: e.g. sterilisation, intrauterine devices (IUD), oral contraceptives, condoms)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2000-02; Primary Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Cumulated headache (intensity x duration) per day based on mean severity per waking hours expressed as area under the curve (AUC) | Day 14 after first drug administration

SECONDARY OUTCOMES:
Proportion of subjects experiencing moderate/severe headache | Day 14 after first drug administration
Proportion of subjects experiencing headache | Day 14 after first drug administration
Cumulated headache (intensity x duration) per day based on maximum severity per day expressed as AUC | Day 14 after first drug administration
Amount of acetylsalicylic acid (ASA) 500 used to cut headache | Day 14 after first drug administration
Changes from baseline in vital signs | Pre-dose and day 17 after first drug administration
Changes from baseline in laboratory tests | Pre-dose and day 17 after first drug administration
Changes from baseline in 12-lead ECG | Pre-dose and day 17 after first drug administration
Changes from baseline in physical examination | Pre-dose and day 17 after first drug administration
Number of patients with adverse events | Up to day 17 after first drug administration